CLINICAL TRIAL: NCT00634686
Title: Effects of Omega-3 Fatty Acids on Bone and Frailty
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Donaghue Medical Research Foundation (Other)
Collaborators: University of Connecticut (Other)
Responsible Party: Anne Kenny, MD, Associate Professor of Medicine, University of Connecticut Center on Aging
Organization: National Institute on Aging (NIA) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AG0096
Record Dates: First submitted 2008-03-11; First posted 2008-03-13 (Estimated); Last update posted 2009-02-02 (Estimated); Status verified 2009-01

CONDITIONS: Osteoporosis; Frailty
Keywords: Omega-3 fatty acids; immune response
MeSH Terms: conditions — Osteoporosis; Frailty | interventions — Calcium; Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Dietary Supplement: DHA/EPA; Dietary Supplement: Calcium with vitamin D
- 2 (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo capsule; Dietary Supplement: Calcium with vitamin D

INTERVENTIONS:
Dietary Supplement: DHA/EPA — 1.2 gram capsule daily for 6 months
  Arms: 1
Dietary Supplement: Placebo capsule — daily for 6 months
  Arms: 2
Dietary Supplement: Calcium with vitamin D — 1000 mg of calcium with 1000 IU vitamin D daily for 6 months

SUMMARY:
The purpose of this study is to examine the effects of essential fatty acid (EFA) supplementation on bone metabolism and frailty in postmenopausal women. The overall hypothesis is that EFA supplementation, via its immunoregulatory and anti-inflammatory activity, will decrease bone turnover, decrease prostaglandins and cytokines associated with bone metabolism and frailty, and change physical outcome measures associated with frailty in postmenopausal women with low bone mass and frailty.

DETAILED DESCRIPTION:
Osteoporosis is a bone thinning disease that results in fractures that occur with minimal trauma. The direct health care costs related to osteoporosis are estimated to be $14 billion per year, comparable to costs in heart failure and asthma. Frailty, or poor physiologic reserve to deal with stressors, is estimated to be 7% in the general population over age 65. The frailty syndrome is characterized by sarcopenia or muscle loss, inflammation, low estrogen, growth hormone and testosterone levels, poor nutrition and disability, and is associated with an increased risk of falls and fracture. Omega-3 fatty acids found in fish oil (eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA)) have been shown to decrease markers of inflammation (cytokines) and decrease death due to heart disease. A number of studies in animals suggest that fish oil (EPA and DHA) supplementation inhibits bone break down, increases calcium absorbed from the diet and enhances calcium in bone. Few studies have assessed the role of n-6 and n-3 fatty acids in the diet in bone disease in humans. As far as we know, no study has evaluated the role of n-3 fatty acids in the frailty syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women over 65 years old
* Spine or hip bone density T score less than -1
* Hand grip strength 2 standard deviations below weight adjusted norms
* Able to travel to the clinical sites for follow-up visits

Exclusion Criteria:

* Any disease that may affect bone metabolism, (i.e Paget's disease, primary hyperparathyroidism)
* Cancer of any kind (except basal or squamous cell of skin) in past 5 years.
* Use of calcitonin, calcitriol, heparin, phenytoin, phenobarbital, and estrogen in the past 6 months
* Use of bisphosphonates, long-term corticosteroids (more than 6 months), methotrexate, or fluoride at any time
* Current use of any medication or herbs with anticoagulant or antiplatelet activity, tetracycline, and magnesium or zinc supplementation
* Estimated creatinine clearance less than 50 ml/min
* History of chronic liver disease or evidence of liver disease on screening
* History of hip fracture or known vertebral fracture within the past year
* Untreated hypertension or a history of clotting disorders
* History of allergy to fish or fish oil

Min Age: 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2007-01; Primary Completion 2009-06 (Estimated); Study Completion 2009-06 (Estimated)

PRIMARY OUTCOMES:
Bone turnover markers | baseline, 3 and 6 months

SECONDARY OUTCOMES:
Bone Mineral Density | baseline, 3 and 6 months
Physical performance measures | baseline, 3 and 6 months
Blood pressure and lab work, including lipids, cytokines, prostaglandins, lymphocyte characterization, and EPA/DHA in blood and plasma | baseline, 3 and 6 months
Cognitive status, mood and depression | baseline, 3 and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Anne Kenny, MD, Principal Investigator — University of Connecticut Center on Aging
Locations (1):
- University of Connecticut Health Center, Farmington, Connecticut, United States

REFERENCES:
- [Background] Arlt W, Callies F, van Vlijmen JC, Koehler I, Reincke M, Bidlingmaier M, Huebler D, Oettel M, Ernst M, Schulte HM, Allolio B. Dehydroepiandrosterone replacement in women with adrenal insufficiency. N Engl J Med. 1999 Sep 30;341(14):1013-20. doi: 10.1056/NEJM199909303411401. PMID 10502590
- [Background] Callies F, Fassnacht M, van Vlijmen JC, Koehler I, Huebler D, Seibel MJ, Arlt W, Allolio B. Dehydroepiandrosterone replacement in women with adrenal insufficiency: effects on body composition, serum leptin, bone turnover, and exercise capacity. J Clin Endocrinol Metab. 2001 May;86(5):1968-72. doi: 10.1210/jcem.86.5.7483. PMID 11344193
- [Background] Morales AJ, Haubrich RH, Hwang JY, Asakura H, Yen SS. The effect of six months treatment with a 100 mg daily dose of dehydroepiandrosterone (DHEA) on circulating sex steroids, body composition and muscle strength in age-advanced men and women. Clin Endocrinol (Oxf). 1998 Oct;49(4):421-32. doi: 10.1046/j.1365-2265.1998.00507.x. PMID 9876338